CLINICAL TRIAL: NCT00543660
Title: Descemet Stripping (Automated) Endothelial Keratoplasty (DSEK or DSAEK)
Acronym: DSAEK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Netherlands Institute for Innovative Ocular Surgery (Other)
Collaborators: Amnitrans Eyebank Rotterdam (Other); Melles CorneaClinic Rotterdam (Unknown)
Responsible Party: Principal Investigator, GRJ Melles, MD, PhD, Director, Netherlands Institute for Innovative Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIIOS.1998.04
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Corneal Dystrophies, Hereditary
Keywords: Corneal transplantation, Descemet membrane, endothelium
MeSH Terms: conditions — Corneal Dystrophies, Hereditary | interventions — Descemet Stripping Endothelial Keratoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention arm DSEK (Experimental): Intervention: DSEK
  Interventions: Procedure: Descemet Stripping Automated Endothelial Keratoplasty (DSAEK)

INTERVENTIONS:
Procedure: Descemet Stripping Automated Endothelial Keratoplasty (DSAEK)
  Other Names: Descemet Stripping Endothelial Keratoplasty (DSEK); Please see www.niios.com

SUMMARY:
To evaluate the transplantation of a posterior corneal disc for the management of corneal endothelial disorders in Descemet Stripping Endothelial Keratoplasty (DSEK) or Descemet Stripping Automated Endothelial Keratoplasty (DSAEK).

DETAILED DESCRIPTION:
Please see above.

ELIGIBILITY:
Inclusion Criteria:

* Corneal endothelial disorders

Exclusion Criteria:

* N/A

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1998-03; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Best spectacle corrected visual acuity | 1998 - 2018

SECONDARY OUTCOMES:
Corneal endothelial cell density | 1998-2018

CONTACTS AND LOCATIONS:
Overall Officials: Gerrit RJ Melles, MD PhD, Principal Investigator — Netherlands Institute for Innovative Ocular Surgery
Locations (1):
- Netherlands Institute for Innovative Ocular Surgery, Rotterdam, Netherlands

REFERENCES:
- [Result] Melles GR. Posterior lamellar keratoplasty: DLEK to DSEK to DMEK. Cornea. 2006 Sep;25(8):879-81. doi: 10.1097/01.ico.0000243962.60392.4f. No abstract available. PMID 17102659